CLINICAL TRIAL: NCT04508270
Title: Physiological Evidence for Early Mobilization in Thoracoscopic Lobectomy
Brief Title: Significance of Early Mobilization After VATS-L
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lin Huang, Medical Doctor, Research fellow, PhD student, Rigshospitalet, Denmark
Other Study IDs: H-20041481
Record Dates: First submitted 2020-07-31; First posted 2020-08-11 (Actual); Last update posted 2020-12-30 (Actual); Status verified 2020-12

CONDITIONS: Lung Neoplasm; Physiology; Exercise; Lung Function; Arterial Oxygen Saturation
Keywords: Postoperative mobilization; Physiology; Thoracoscopy; Lobectomy
MeSH Terms: conditions — Lung Neoplasms; Motor Activity | interventions — Early Ambulation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Early mobilization — Mobilization as soon as patients can, which is not limited on walking

SUMMARY:
The main endpoint is physiological rehabilitation after VATS-L under early mobilization. The secondary endpoints are exploring the effect of early mobilization on postoperative physiology.

Investigators hypothesis that early mobilization is clearly advantaged to advance the physiological recovery.

ELIGIBILITY:
Inclusion Criteria:

1. VATS lobectomy;
2. Speak and understand Danish or English;
3. Informed consent obtained.

Exclusion Criteria:

1. Co-VATS lobectomy (more than one lobe resection);
2. Supplementary oxygen therapy later 6 h after surgery;
3. No willing to wear electronic device;
4. No willing to exam arterial oxygen saturation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for VATS-L.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2020-09-08 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Postoperative forced expiratory volume in one second (FEV1) | Through study completion, an average of 3 days
  FEV1 is the amount of air you can force from your lungs in one second. Participants will be examed via spirometer.
Postoperative arterial oxygen saturation. | Through study completion, an average of 3 days
  Oxygen saturation is the fraction of oxygen-saturated hemoglobin relative to total hemoglobin (unsaturated + saturated) in the blood. Participants will be tested via oximeter.

SECONDARY OUTCOMES:
The quantization of activity counts | Through study completion, an average of 3 days
The quantization of pain | Through study completion, an average of 3 days
  The numeric rating scale (NRS) ranging from 0 (no pain) to 10 (excruciating pain) is used to score postoperative pain.
length of stay in hospital | Through study completion, an average of 3 days
Duration of chest tube | Through study completion, an average of 2 days
Postoperative complications | up to 30 days
  Pneumothorax, subcutaneous emphysema, pneumonia, empyema, bleeding, pulmonary embolism, prolong air leakage, re-intervention, re-surgery and re-admission will be recording specifically.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Huang, MD, Principal Investigator — Rigshospitalet, Denmark; Henrik Kehlet, Professor, MD, DMSc, Study Director — Rigshospitalet, Denmark; Rene H Petersen, Professor, MD, PhD, Study Chair — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Background] Ljungqvist O, Scott M, Fearon KC. Enhanced Recovery After Surgery: A Review. JAMA Surg. 2017 Mar 1;152(3):292-298. doi: 10.1001/jamasurg.2016.4952. PMID 28097305
- [Background] Kehlet H. Multimodal approach to control postoperative pathophysiology and rehabilitation. Br J Anaesth. 1997 May;78(5):606-17. doi: 10.1093/bja/78.5.606. PMID 9175983
- [Background] Batchelor TJP, Rasburn NJ, Abdelnour-Berchtold E, Brunelli A, Cerfolio RJ, Gonzalez M, Ljungqvist O, Petersen RH, Popescu WM, Slinger PD, Naidu B. Guidelines for enhanced recovery after lung surgery: recommendations of the Enhanced Recovery After Surgery (ERAS(R)) Society and the European Society of Thoracic Surgeons (ESTS). Eur J Cardiothorac Surg. 2019 Jan 1;55(1):91-115. doi: 10.1093/ejcts/ezy301. PMID 30304509
- [Background] Haines KJ, Skinner EH, Berney S; Austin Health POST Study Investigators. Association of postoperative pulmonary complications with delayed mobilisation following major abdominal surgery: an observational cohort study. Physiotherapy. 2013 Jun;99(2):119-25. doi: 10.1016/j.physio.2012.05.013. Epub 2012 Sep 23. PMID 23219632
- [Background] Mynster T, Jensen LM, Jensen FG, Kehlet H, Rosenberg J. The effect of posture on late postoperative oxygenation. Anaesthesia. 1996 Mar;51(3):225-7. doi: 10.1111/j.1365-2044.1996.tb13637.x. PMID 8712320
- [Background] Hanada M, Kanetaka K, Hidaka S, Taniguchi K, Oikawa M, Sato S, Eguchi S, Kozu R. Effect of early mobilization on postoperative pulmonary complications in patients undergoing video-assisted thoracoscopic surgery on the esophagus. Esophagus. 2018 Apr;15(2):69-74. doi: 10.1007/s10388-017-0600-x. Epub 2017 Dec 16. PMID 29892929
- [Background] Liu Z, Tao X, Chen Y, Fan Z, Li Y. Bed rest versus early ambulation with standard anticoagulation in the management of deep vein thrombosis: a meta-analysis. PLoS One. 2015 Apr 10;10(4):e0121388. doi: 10.1371/journal.pone.0121388. eCollection 2015. PMID 25860350
- [Background] Ueda K, Sudoh M, Jinbo M, Li TS, Suga K, Hamano K. Physiological rehabilitation after video-assisted lung lobectomy for cancer: a prospective study of measuring daily exercise and oxygenation capacity. Eur J Cardiothorac Surg. 2006 Sep;30(3):533-7. doi: 10.1016/j.ejcts.2006.05.025. Epub 2006 Jul 20. PMID 16857371
- [Background] Rogers LJ, Bleetman D, Messenger DE, Joshi NA, Wood L, Rasburn NJ, Batchelor TJP. The impact of enhanced recovery after surgery (ERAS) protocol compliance on morbidity from resection for primary lung cancer. J Thorac Cardiovasc Surg. 2018 Apr;155(4):1843-1852. doi: 10.1016/j.jtcvs.2017.10.151. Epub 2017 Dec 19. PMID 29352586
- [Background] Chang NW, Lin KC, Lee SC, Chan JY, Lee YH, Wang KY. Effects of an early postoperative walking exercise programme on health status in lung cancer patients recovering from lung lobectomy. J Clin Nurs. 2014 Dec;23(23-24):3391-402. doi: 10.1111/jocn.12584. Epub 2014 Mar 20. PMID 24646333
- [Background] Kirkeby-Garstad I, Wisloff U, Skogvoll E, Stolen T, Tjonna AE, Stenseth R, Sellevold OF. The marked reduction in mixed venous oxygen saturation during early mobilization after cardiac surgery: the effect of posture or exercise? Anesth Analg. 2006 Jun;102(6):1609-16. doi: 10.1213/01.ANE.0000219589.03633.BF. PMID 16717296
- [Derived] Huang L, Kehlet H, Petersen RH. Effect of posture on pulmonary function and oxygenation after fast-tracking video-assisted thoracoscopic surgery (VATS) lobectomy: a prospective pilot study. Perioper Med (Lond). 2021 Sep 2;10(1):26. doi: 10.1186/s13741-021-00199-z. PMID 34470657